CLINICAL TRIAL: NCT03031301
Title: A Prospective, Multicenter, Randomized, Double-blind, Sham-controlled Study to Assess the Efficacy and Safety of the Vibrant Capsule Administered 5 Times Per Week
Brief Title: A Study to Assess the Efficacy and Safety of the Vibrant Capsule Administered 5 Times Per Week
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vibrant Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 240CLD
Record Dates: First submitted 2017-01-16; First posted 2017-01-25 (Estimated); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2019-01

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Vibrant capsule (Active Comparator): Patients will receive the Vibrant capsule 5 times a week for 8 weeks of treatment
  Interventions: Device: Vibrant capsule
- Sham capsule (Sham Comparator): Patients will receive the sham capsule (activated, non-vibrating) 5 times a week for 8 weeks of treatment
  Interventions: Device: Sham capsule

INTERVENTIONS:
Device: Vibrant capsule — One Vibrant capsule will be ingested 5 times per week for 8 weeks of treatment.
  Arms: Vibrant capsule
Device: Sham capsule — One Sham capsule will be ingested 5 times per week for 8 weeks of treatment.
  Arms: Sham capsule

SUMMARY:
The study is a prospective, adaptive, multicenter, randomized, double-blind, Sham-controlled study, to evaluate the efficacy and safety of the Vibrant Capsule in relieving constipation in subjects with functional constipation.

Two arms will be assessed:

* Vibrant Capsule administered 5 times per week
* Sham Capsule administered 5 times per week

DETAILED DESCRIPTION:
The study is a prospective, adaptive, multicenter, randomized, double-blind, Sham-controlled study, to evaluate the efficacy and safety of the Vibrant Capsule in relieving constipation in subjects with functional constipation.

Two arms will be assessed:

* Vibrant Capsule administered 5 times per week
* Sham Capsule administered 5 times per week

Subjects will follow a 2 weeks baseline period and then take the Vibrant Capsule for a treatment period of 8 weeks.

Data reporting will be done on an electronic Case Report Form (eCRF) and an eDiary.

Subjects will be asked to refrain from taking any medication or supplement to relieve their constipation, during the entire study period.

After the 14 days of run-in period, the subjects will return and eligibility will be re-assessed. Subjects will be trained on how to use the base unit and will swallow the first capsule on site the day of baseline visit. They will activate and ingest the rest of the capsules at home by themselves, using the base unit.

Subjects will be instructed to complete a simple subject eDiary each day throughout the duration of the study. A final visit will take place at the end of the 8 week treatment period.

Subjects will receive phone calls at least once a week and subject compliance will be monitored during the 8 weeks of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 22 years and older
2. Subjects with Chronic Idiopathic Constipation (CIC) according to Rome III criteria and who have not experienced relief of their symptoms from available therapies
3. Subjects with an average of <3 Spontaneous Bowel Movements (SBM) per week and ≥1 SBM per week
4. Normal colonoscopy performed within 10 years prior to study participation, unless the subjects are <50 years old and without alarm signs and/or symptoms
5. Subject signed the Informed Consent Form (ICF)
6. Female subjects must have a negative pregnancy test

Exclusion Criteria:

1. History of complicated/obstructive diverticular disease
2. History of intestinal or colonic obstruction, or suspected intestinal obstruction.
3. History of significant gastrointestinal disorder, including any form of inflammatory bowel disease or gastrointestinal malignancy (celiac disease is accepted if the subject has been treated and is in remission)
4. History of gastroparesis
5. Use of any of the following medications:

   * Medications that may affect intestinal motility, prokinetics, anti-depressants, anti-Parkinsonian medications, opiates, opioids, calcium-channel blockers, aluminum/magnesium hydroxide
   * With the exception of antidepressants, thyroid or hormonal replacement therapy, when the subject has been on a stable dose for at least 3 months prior to enrollment.
6. Clinical evidence of significant respiratory, cardiovascular, renal, hepatic, biliary, endocrine, psychiatric or neurologic disease.
7. Presence of cardiac pacemaker or gastric electrical stimulator.
8. History of, or current eating disorders, such as anorexia, bulimia, or compulsory overeating.
9. Diagnosis of mega-rectum or colon, congenital anorectal malformation, clinically significant rectocele, history of intestinal resection (with an exception for appendectomy, cholecystectomy and inguinal hernia repair), history of bariatric surgery or evidence of any structural abnormality of the gastrointestinal tract that might affect transit
10. History of Zenker's diverticulum, dysphagia, Barrett's esophagus, esophageal stricture or achalasia
11. Chronic use of non-steroidal anti-inflammatory drugs (NSAIDs)
12. Subjects with pelvic floor dysfunction/defecatory disorder
13. Participation in another clinical study within one month prior to screening.
14. Women who are pregnant or lactating

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dvora Darky, Study Director — Vibrant Ltd.
Locations (2):
- United States (2):
  - Avant Guntersville, Guntersville, Alabama
  - Floridian Research Institute, Miami, Florida

IPD SHARING:
Plan to Share IPD: No
Data from this study will be presented in future Vibrantgastro publications.

REFERENCES:
- [Derived] Rao SSC, Lembo A, Chey WD, Friedenberg K, Quigley EMM. Effects of the vibrating capsule on colonic circadian rhythm and bowel symptoms in chronic idiopathic constipation. Neurogastroenterol Motil. 2020 Nov;32(11):e13890. doi: 10.1111/nmo.13890. Epub 2020 May 25. PMID 32449277

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vibrant Capsule | Sham Capsule
Started | 89 | 93
Completed | 71 | 65
Not Completed | 18 | 28
Not completed — Protocol Violation | 4 | 8
Not completed — Withdrawal by Subject | 7 | 4
Not completed — Lost to Follow-up | 4 | 12
Not completed — Noncompliance | 1 | 3
Not completed — Technical issue | 1 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vibrant Capsule | Sham Capsule | Total
Number analyzed (Participants) | 89 | 93 | 182
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.36 (13.08) | 42.67 (11.16) | 43.99 (12.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 71 | 142
  Male | 18 | 22 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 37 | 29 | 66
  Hispanic or Latino | 17 | 22 | 39
  Black or African American | 32 | 33 | 65
  Native or Indian American | 1 | 4 | 5
  Asian/ Pacific Islander | 1 | 3 | 4
  Other | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 89 | 93 | 182
Duration of constipation [Mean (Standard Deviation); unit: years] | 11.67 (12.46) | 13.09 (12.19) | 12.40 (12.31)

OUTCOME MEASURES:

1. Primary Outcome: CSBM1- Number of Participants With an Increase of at Least One Weekly Complete Spontaneous Bowel Movement (CSBM) During at Least 6 of the 8 Weeks of Treatment
Description: CSBM1 success rate, defined as an increase from the run-in period of at least one weekly Complete Spontaneous Bowel Movement (CSBM) during at least 6 of the 8 weeks of treatment
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Vibrant Capsule | Sham Capsule
Number analyzed (Participants) | 89 | 93
Participants | 24 | 33

2. Primary Outcome: CSBM2- Number of Participants With an Increase of at Least 2 Weekly Complete Spontaneous Bowel Movement (CSBM) During at Least 6 of the 8 Weeks of Treatment
Description: CSBM2 success rate, defined as an increase from the run-in period of at least 2 weekly Complete Spontaneous Bowel Movement (CSBM) during at least 6 of the 8 weeks of treatment
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Vibrant Capsule | Sham Capsule
Number analyzed (Participants) | 89 | 93
Participants | 16 | 26

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Vibrant Capsule | Sham Capsule
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/93
Serious Adverse Events (participants affected / at risk) | 1/89 | 1/93
Other Adverse Events (participants affected / at risk) | 28/89 | 19/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vibrant Capsule (N=89) | Sham Capsule (N=93)
Traumatic Fracture Of Pelvis (Musculoskeletal and connective tissue disorders) | 1 | 0 — Traumatic Fracture Of Pelvis, not related to the device
Anxiety Attack (Psychiatric disorders) | 0 | 1 — Anxiety Attack, not related to the device
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vibrant Capsule (N=89) | Sham Capsule (N=93)
Nausea (Gastrointestinal disorders) | 7 (8) | 2 (2) — Nausea
Sensation of vibration (Product Issues) | 15 (30) | 2 (2) — Sensation of vibration
Bloating (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal Cramping (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Decrease In The Frequency In Bm (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Extreme Lower Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal Bleeding (Gastrointestinal disorders) | 1 (1) | 1 (1)
Uncomfortable Bm (Gastrointestinal disorders) | 0 (0) | 1 (1)
Viral Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Permission to use study data is required

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-06): https://cdn.clinicaltrials.gov/large-docs/01/NCT03031301/Prot_SAP_000.pdf